CLINICAL TRIAL: NCT06689267
Title: Initial CT Perfusion-Guided Strategy Versus Invasive Coronary Angiography in Patients With Suspected Non-ST-Segment Elevation Myocardial Infarction
Brief Title: Initial CT Perfusion-Guided Strategy for Suspected NSTEMI
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, Director of the Department of Cardiology, Professor, Academician of the Chinese Academy of Sciences., Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ZS-SMART
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-11

CONDITIONS: Non-ST Elevation Myocardial Infarction
Keywords: NSTEMI; CT angiography; CT perfusion; invasive angiography
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial CT perfusion (Experimental): Patients enrolled in the Initial CT perfusion group will first undergo CTA and CTP examinations. Based on the results of these tests, the treatment team will then decide whether to proceed with conservative medical therapy or perform coronary angiography.
  Interventions: Diagnostic Test: computed tomography myocardial perfusion
- Invasive Coronary Angiography (Active Comparator): Patients enrolled in the Invasive Coronary Angiography group will directly undergo coronary angiography. If necessary, intracoronary imaging (including IVUS and OCT) will be performed. Based on the results of these tests, the treatment team will then decide whether to proceed with conservative medical therapy or interventional treatment (including stent implantation or balloon angioplasty).
  Interventions: Procedure: Invasive Coronary Angiography

INTERVENTIONS:
Diagnostic Test: computed tomography myocardial perfusion — The diagnostic value of CT perfusion (CTP) has been established in patients with stable coronary artery disease, but relevant studies have not yet been conducted in suspected NSTEMI patients. This study aims to explore the diagnostic and therapeutic value of an initial CTP strategy for suspected NSTEMI patients.
  Arms: Initial CT perfusion
Procedure: Invasive Coronary Angiography — Patients enrolled in the Invasive Coronary Angiography group will directly undergo coronary angiography. If necessary, intracoronary imaging (including IVUS and OCT) will be performed.
  Arms: Invasive Coronary Angiography

SUMMARY:
Non-ST elevation myocardial infarction (NSTEMI) is a relatively complex type of myocardial infarction, characterized by chest pain symptoms and elevated troponin levels. However, some patients initially diagnosed with suspected NSTEMI are found not to have severe stenosis upon coronary angiography. Recent studies have shown that initial imaging examinations (including CTA and CMR) in suspected NSTEMI patients can help reduce the need for coronary angiography. The diagnostic value of CT perfusion (CTP) has been established in patients with stable coronary artery disease, but relevant studies have not yet been conducted in suspected NSTEMI patients. This study aims to explore the diagnostic and therapeutic value of an initial CTP strategy for suspected NSTEMI patients. Additionally, we will conduct a cardiovascular health questionnaire to investigate the impact and prognostic value of factors such as adverse lifestyle and inflammation levels in these patients.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is caused by acute and persistent ischemia and hypoxia of the coronary arteries, leading to myocardial necrosis. Clinically, it often presents as severe and prolonged retrosternal pain, accompanied by elevated serum myocardial enzyme levels and progressive changes in the electrocardiogram (ECG). Complications may include arrhythmias, shock, or heart failure, which can be life-threatening.

Non-ST elevation myocardial infarction (NSTEMI) is a more complex type of AMI. It presents with chest pain and elevated troponin levels, but without clear ischemic changes on the ECG, making clinical diagnosis challenging. Additionally, NSTEMI patients are highly heterogeneous, influenced by factors like lifestyle and inflammation. Current clinical guidelines recommend coronary angiography for these patients. However, previous studies have shown that approximately one-third of suspected NSTEMI patients do not exhibit significant coronary stenosis on angiography. Minimizing unnecessary invasive coronary angiography for such patients has become a pressing issue.

Recent clinical studies have explored the value of initial imaging tests in guiding treatment strategies for NSTEMI patients. The CARMENTA study found that performing CTA or MRI as the first-line test in suspected NSTEMI patients could reduce the need for subsequent invasive coronary angiography by 13% and 34%, respectively, and improve the positive detection rate on later angiography. The OxAMI study also showed that in patients with suspected NSTEMI who underwent MRI, only 67% had myocardial infarction, and even among those who subsequently underwent angiography and were found to have severe stenosis, CMR indicated infarction in only 84%. These findings suggest that while CTA can help rule out some myocardial infarction cases, its diagnostic value in suspected NSTEMI remains limited.

With advances in imaging technology, CT myocardial perfusion (CTP) has shown potential in more accurately identifying ischemic myocardium in coronary artery disease patients, thereby enhancing the diagnostic power of CTA. However, the diagnostic value of CTP for suspected NSTEMI patients remains unclear. Furthermore, technology now allows for simultaneous CTA and CTP testing without significantly increasing radiation exposure. This combined approach offers promise for more accurate diagnosis in suspected NSTEMI patients without a marked increase in radiation dose.

Therefore, this study aims to investigate the diagnostic and therapeutic value of an initial CTP strategy in suspected NSTEMI patients. Additionally, we will conduct a cardiovascular health questionnaire survey to explore the impact and prognostic value of adverse lifestyle factors and inflammation levels in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stable chest tightness or chest pain, aged ≥18 years
2. No ST elevation or dynamic ST-T changes on the ECG
3. Elevated TNT (greater than 14 ng/L three hours after symptom onset)

Exclusion Criteria:

1. Persistent chest pain or ECG indicating dynamic ST-T changes,
2. Hemodynamic instability
3. Known history of coronary artery disease
4. Contraindications for CT perfusion or coronary angiography
5. Coexisting conditions such as pregnancy, cancer, severe valvular heart disease, or liver/kidney dysfunction
6. Other diseases with a life expectancy of less than one year
7. Inability to sign informed consent or, in the researcher's judgment, poor compliance, making it unlikely the patient can complete the study as required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who ultimately undergo coronary angiography. | From enrollment to 1 week or at the time of discharge from hospital, whichever came first
  Patients enrolled in the Initial CT perfusion group will first undergo CTA and CTP examinations. Based on the results of these tests, the treatment team will then decide whether to proceed with conservative medical therapy or coronary angiography. According to previous research data, approximately 20-30% of patients will not require coronary angiography. In contrast, patients enrolled in the Invasive Coronary Angiography group will undergo coronary angiography in 100% of cases.

SECONDARY OUTCOMES:
MACE | From enrollment to the follow-up of 1 year
  MACE was a composite of all- cause mortality, recurrent MI, unplanned coronary revascularization after the index event, or congestive heart failure requiring hospitalization.

OTHER OUTCOMES:
Perioperative adverse events | From enrollment to the follow-up of 1 year
  adverse events including significant bleeding, contrast-induced nephropathy, renal failure, nephrogenic systemic fibrosis, allergic reaction requiring urgent therapy, dissection or perforation of a vessel, stroke, or transient ischemic attack

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No